CLINICAL TRIAL: NCT00565929
Title: MVA-BN (IMVAMUNE®) Immunization in Persons Who Have Undergone Prior Hematopoietic Stem Cell Transplant (HSCT): A Phase I, Placebo-Controlled Study of the Safety, Reactogenicity and Immunogenicity of MVA Immunization
Brief Title: Safety, Reactogenicity and Immunogenicity of MVA in Hematopoietic Stem Cell Transplant (HSCT) Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-0042; 5U54AI057159-10 (NIH)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2012-09

CONDITIONS: Variola Major (Smallpox)
Keywords: Variola major, smallpox, vaccine, hematopoietic stem cell transplant
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group A: MVA-BN 1 X 10^7 TCID 50 (Experimental): 10 participants to receive vaccine dose 1X10^7 TCID 50; 2 participants to receive placebo.
  Interventions: Drug: Placebo; Biological: MVA-BN
- Group B: MVA-BN 1 X 10^8 TCID 50 (Experimental): 10 participants to receive vaccine dose 1X10^8 TCID 50; 2 participants to receive placebo.
  Interventions: Drug: Placebo; Biological: MVA-BN

INTERVENTIONS:
Drug: Placebo — Sterile saline (0.9%).
Biological: MVA-BN — The smallpox vaccine is a liquid frozen solution formulated to contain 0.605 mg Tris and 4.090 mg sodium chloride (NaCl) per 0.5 mL dose. The concentration of the virus will be 1 X 10^8 tissue culture infectious dose 50 (TCID 50) per 0.5 mL dose and may be diluted in a solution of 0.9% saline prior to vaccination. Smallpox vaccine administered in 2 doses approximately 28 days apart in one of the following doses: 1X10^7 or 1X10^8 TCID 50.

SUMMARY:
The purpose of this study is to compare how the body's immune system reacts to a vaccine against smallpox infection, called Modified Vaccinia Ankara (MVA) and to evaluate the safety of this vaccine. Study participants will include 24 adults, ages 18-60 years, who have undergone a stem cell transplant more than 2 years ago. Study procedures will include a physical exam, blood samples, heart activity assessments, and urine samples. Participants will be assigned to 1 of 2 possible study vaccine groups. The participants will receive 1 of 2 possible vaccine doses or placebo (substance containing no medication) 28 days apart. Participants will make at least 8 visits to the clinic during the course of the study; additional visits may be needed if the participant experiences side effects from the vaccine. Participants may be involved in study related procedures for about 6 months.

DETAILED DESCRIPTION:
In the event of a smallpox outbreak, or threat of one, mass immunization of all vulnerable individuals would take place. This would include persons with immunodeficiency as seen post Hematopoietic Stem Cell Transplant (HSCT). The current Food and Drug Administration (FDA) approved smallpox vaccine (Dryvax®) is a live replicating virus (vaccinia) and is contraindicated in both immunocompromised persons and those in close physical contact with them. The Modified Vaccinia Ankara (MVA), specifically IMVAMUNE® has been developed as a safer, less reactogenic vaccine against smallpox. Study participants will include 24 male or female participants, from 18 to 60 years of age. This study assesses the safety, reactogenicity and immunogenicity of 2 doses of MVA-BN (IMVAMUNE®) given to persons who have undergone an HSCT more than 2 years prior to study participation. There are 2 arms in the study, each receiving 2 doses 28 days apart of either 1 x 10^7 or 1 x 10^8 tissue culture infectious dose 50 (TCID50). Each arm will be comprised of 12 subjects, 10 of whom will receive IMVAMUNE® and 2 of whom will receive placebo under a double blind, randomized allocation. Subjects will be followed for safety and reactogenicity. Clinical assessments will be performed and blood samples will be obtained sequentially for safety and immunogenicity determinations. All subjects will complete a memory aid for 15 days after each vaccination to record oral temperature and note the occurrence of solicited and unsolicited adverse events as well as any medication use. Adverse events will be collected for 56 days after each vaccination. Serious adverse events and concomitant medications will be collected throughout the entire study period. Study staff will assess subjects clinically at days 14 and 28 after each vaccination and on days 42, 56, 84, and 180. Hematology and blood chemistry studies including hemoglobin, white blood cell and platelet counts and kidney and liver function tests will be obtained. Electrocardiogram and Troponin I or T will be obtained prior to first vaccination and on days 14 and 28 after each immunization and at day 180. Clinical laboratory assays will be conducted in the clinical laboratory at both the Brigham and Women's Hospital or the Dana Farber Cancer Institute. The primary objective of this study is to determine the safety and reactogenicity of MVA in persons who have undergone allogeneic HSCT more than 2 years prior to study participation. The secondary objective of this study is to determine the immunogenicity of MVA in persons who have undergone HSCT more than 2 years prior to study participation. Immunogenicity will be determined by humoral immune responses and cell mediated immune responses.

ELIGIBILITY:
Inclusion Criteria:

General:

* Age: 18 to 60
* Complete a written assessment of understanding prior to enrollment and verbalize understanding of all questions answered incorrectly
* Informed consent: Be able, willing, and have signed the informed consent form
* Undergone stem cell transplant more than 2 years prior to enrollment
* Current Health: Be in good general health without evidence of active malignancy and off immunosuppressant medications. Without evidence of clinically significant medical history, physical examination findings, or clinically significant abnormal laboratory results. A clinically significant condition or process includes one or more of the following:

  1. An active condition that is life threatening
  2. A condition for which repeated injections or blood draws may pose additional risk to the participant
  3. A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being
  4. A condition or process in which signs or symptoms could be confused with reactions to vaccine

Laboratory:

* Hematology and chemistries: Chemistries within 1.25x of the institutional normal limits for age and sex for alanine aminotransferase (ALT), aspartate aminotransferase (AST), Alkaline Phos, and Total Bilirubin. Creatinine less than or equal to 1.8 mg/dL. Platelets and Troponin I or T must be within normal range. Hemoglobin above 10.5 gm/dL for women and 11.5 gm/dL for men and white blood cells (WBC) between 3,000 and 12,500 cells/mm^3.
* Negative for Hepatitis B surface antigen and Hepatitis C virus (HCV) antibodies (If HCV antibodies are positive, and negative for HCV by polymerase chain reaction (PCR), subject is eligible)
* Negative Food and Drug Administration (FDA)-approved human immunodeficiency virus (HIV) blood test within 8 weeks prior to enrollment
* Normal urine dipstick or urinalysis:

  1. Negative glucose, and
  2. Negative or trace protein and negative or trace hemoglobin (if trace hemoglobin is present, a urinalysis is required to exclude participants with counts greater than the institutional normal range)

In addition to meeting ALL of the above criteria, FEMALE participants must meet BOTH of the following criteria:

* Negative serum or urine Beta-human chorionic gonadotropin (HCG) pregnancy test performed within 24 hours prior to any vaccination
* Reproductive status: A female participant either must:

  1. not be of reproductive potential (Reproductive potential in women is defined as not having reached menopause (no menses for one year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation.)
  2. be with a male partner(s) throughout the duration of the study who has undergone successful vasectomy (A vasectomy is considered successful if a woman reports that a male partner has (1) microscopic documentation of azospermia, or (2) a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy), or
  3. agree to avoid pregnancy through alternative methods and agree to consistently use contraception for at least 21 days prior to enrollment until 1 month after last vaccination. Contraception is defined as using one of the following methods: condoms (male or female with or without a spermicide), diaphragm or cervical cap with spermicide, intrauterine device (IUD), or hormone-based therapy, e.g., contraceptive pills, Norplant, or Depo-Provera.

Exclusion Criteria:

* Chronic Graft versus Host Disease (GVHD) requiring systemic immunosuppressive medication within the last 6 months.
* Immunosuppressive medications within 30 days prior to initial study vaccine administration, e.g., oral/parenteral corticosteroids, and/or cytotoxic medications. Not excluded: A participant using any of the following is not excluded: corticosteroid nasal spray for allergic rhinitis; or topical corticosteroids as prescribed by a physician for an acute, uncomplicated dermatitis; or over the counter medications (including topical corticosteroids for an acute, uncomplicated dermatitis); use of rapidly tapered steroids for an acute isolated condition, excluding asthma which is addressed separately-within 28 days prior to vaccine administration.
* Asthma that is unstable, e.g., use of oral or intravenous corticosteroids, hospitalization or intubation during the past 2 years.

  a. In addition, exclude a participant who routinely uses a moderate to high dose inhaled corticosteroids (e.g., more than equivalent of 264 micrograms (mcg) fluticasone; 600 mcg budesonide; 240 mcg beclomethasone; 1000 mcg flunisolide, 750 mcg triamcinolone or 200 mcg mometasone, as a daily dose).
* Receipt of immunoglobulin within 60 days prior to initial study vaccine administration.
* Receipt of live attenuated vaccines within 30 days prior to initial study vaccine administration.
* Receipt of medically indicated subunit or killed vaccines, e.g., influenza, pneumococcal, or allergy treatment with antigen injections within 14 days prior to initial study vaccine administration.
* Participant has a history of any of the following:

  1. Acute febrile illness on the day of vaccination
  2. Eczema or atopic dermatitis (past or present)
  3. Acute skin disorders of large magnitude (greater than 2x2 cm), e.g., burns or lacerations
  4. History or presence of skin cancer at vaccination site(s)
  5. Heart disease including history of a myocardial infarction (MI), angina, congestive heart failure (CHF), or pericardial pathology
  6. Twenty percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp).
* Known allergy to eggs.
* History of serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. Not excluded: A participant who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Bleeding disorder diagnosed by a doctor and that is clinically active, e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions. Not excluded: A participant who states he/she has easy bruising or bleeding, but does not carry a formal diagnosis, and has had intramuscular (IM) injections and blood draws without any adverse experience, is not excluded.
* Active Seizure disorder. Not excluded: A participant with a history of a seizure disorder whose last seizure was over 1 year ago.
* Psychiatric condition that precludes compliance with the protocol.
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or a participant's ability to give informed consent.
* Female participants: Participant is pregnant and or breast-feeding.
* Currently taking investigational agents. Not excluded: participation in a study where the participant is not receiving an investigational agent or the participant is in the follow up phase of a study and the investigational agent was given more than 3 months prior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety: acute reactogenicity, both local and systemic; and hematologic and clinical chemistry laboratory values. | Day 0-180.

SECONDARY OUTCOMES:
Immunogenicity: humoral and cell-mediated immune responses. | Screening, Days 14 and 28 after 1st vaccination; Days 0, 14, 28, 56, and 152 after 2nd vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital - Infectious Diseases, Boston, Massachusetts, United States

REFERENCES:
- [Result] Walsh SR, Wilck MB, Dominguez DJ, Zablowsky E, Bajimaya S, Gagne LS, Verrill KA, Kleinjan JA, Patel A, Zhang Y, Hill H, Acharyya A, Fisher DC, Antin JH, Seaman MS, Dolin R, Baden LR. Safety and immunogenicity of modified vaccinia Ankara in hematopoietic stem cell transplant recipients: a randomized, controlled trial. J Infect Dis. 2013 Jun 15;207(12):1888-97. doi: 10.1093/infdis/jit105. Epub 2013 Mar 12. PMID 23482644